CLINICAL TRIAL: NCT04832750
Title: Depression-Reduction by Accelerated Personalized NeuroModulation and Its Effects on Sleep
Acronym: DREAMS
Status: Completed | Type: Observational
Sponsor: University of Oldenburg (Other)
Collaborators: Marc Onken, M.Sc. (Unknown); Christina Mueller, M.Sc. (Unknown)
Responsible Party: Principal Investigator, Dirk Scheele, Deputy Lab Head, University of Oldenburg
Other Study IDs: DREAMS
Record Dates: First submitted 2021-03-26; First posted 2021-04-06 (Actual); Last update posted 2024-12-11 (Actual); Status verified 2024-12

CONDITIONS: Major Depressive Episode; Major Depressive Disorder; Borderline Personality Disorder
Keywords: rTMS; Theta Burst Stimulation; Neuronavigation; Major Depressive Episode; Borderline Personality Disorder; Sleep; Interoception; Cognitive Control; fMRI
MeSH Terms: conditions — Depressive Disorder, Major; Borderline Personality Disorder

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Weeks
Biospecimen Retention: Samples Without DNA — Blood samples without DNA analysis Saliva samples without DNA analysis
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (3):
- Major Depressive Episode: At least one failed pharmaco trial in current episode
  Interventions: Device: intermittent theta burst stimulation (iTBS) or sham stimulation
- Major Depressive Episode with comorbid Borderline Personality Disorder: At least one failed pharmaco trial in current episode
  Interventions: Device: intermittent theta burst stimulation (iTBS) or sham stimulation
- Healthy Controls: No psychiatric disorders

INTERVENTIONS:
Device: intermittent theta burst stimulation (iTBS) or sham stimulation — 30 sessions of iTBS over 2 weeks (3 sessions per day, 5 days per week)
  Groups: Major Depressive Episode; Major Depressive Episode with comorbid Borderline Personality Disorder

SUMMARY:
Advances in repetitive transcranial magnetic stimulation (rTMS) protocols with intermittent theta-burst stimulation (iTBS) have significantly decreased the duration for one single session and thereby enabled accelerated treatment plans with multiple sessions per day, potentially reducing the total treatment duration. This randomized, placebo-controlled study investigates the effects of accelerated iTBS treatment with connectivity-informed neuronavigation on symptom severity, sleep, interoception, and cognitive control in patients with major depressive disorder and with or without comorbid borderline personality disorder using magnetic resonance imaging (MRI).

DETAILED DESCRIPTION:
Repetitive transcranial magnetic stimulation (rTMS) is a safe and efficacious treatment option for treatment-resistant depression. Advances in rTMS protocols with intermittent theta-burst stimulation (iTBS) have significantly decreased the duration for one single session and thereby enabled accelerated treatment plans with multiple sessions per day, potentially reducing the total treatment duration. Major depressive disorder (MDD) is characterized by impairments in various domains including sleep, impulse control, and interoception. Borderline personality disorder (BPD) is characterized by fear of abandonment, mood swings, and an unstable perception of self and often occurs with comorbid MDD. This comorbidity frequently impedes treatment of the BPD.

In this randomized, placebo-controlled study, 60 patients with treatment-resistant MDD (30 verum group, 30 sham group) and 60 patients with treatment-resistant MDD and comorbid BPD (30 verum group, 30 sham group) will receive two weeks of connectivity-informed iTBS of the left dorsolateral prefrontal cortex (DLPFC; 3 sessions per day, 5 days per week). Before and after the treatment phase, (functional) magnetic resonance imaging (fMRI) will be performed. The effects of iTBS will be tested in four domains: (1) symptom severity (MDD and BPD symptoms), (2) sleep quality (sleep questionnaires and various sleep parameters monitored via an electroencephalography (EEG) headband), (3) neurocognitive effects (vigilance and response inhibition measured with behavioral and fMRI tasks), and (4) interoception (interoceptive attention measured with behavioral and fMRI tasks). Furthermore, before the start of the two-weeks treatment, a single iTBS session ("forecaster session") will be conducted to explore the validity of early symptom/mood responses and hormonal changes for the prediction of the the treatment outcome. Treatment effects will be analyzed within and across patient groups (MDD and MDD + BPD). In addition, domain-specific treatment effects will be analyzed as a function of distinct iTBS targets within the DLPFC.To evaluate pathological biases, the investigators will compare the patients' data with a control group of 30 healthy participants who will also be tested twice (without iTBS).

ELIGIBILITY:
Inclusion Criteria:

* Participant is able to provide consent.
* Diagnosis of major depressive disorder (MDD) according to DSM-V criteria.
* During the current episode, treatment-resistant MDD (at least one failed pharmacological trial of adequate dose and duration)
* For the MDD group with comorbid borderline personality disorder (BPD): diagnosis of BPD according to the Diagnotic Statistical Manual V (DSM-V) criteria.
* For healthy controls: no psychiatric or neurological illness.

Exclusion Criteria:

* For the MDD group without BPD: BPD diagnosis
* The participant does not fulfill requirements for iTBS treatment according to safety guidelines.
* The participant does not fulfill requirements for MRI measurements according to safety guidelines.
* Pregnancy or breast-feeding.
* Acute suicidality.
* Neurological illness (e.g. dementia, Parkinson's disease, chorea huntington, multiple sclerosis).
* increased current risk for epileptic seizure.
* comorbid diagnosis of schizophrenia or psychotic symptoms, bipolar disorder, and substance use disorder within the last 6 months.
* Conditions related to increased intracranial pressure.
* Brain injury or stroke.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients at the Department of Psychiatry, University of Oldenburg. The patients' diagnosis of MDD and BPD will be verified via the structured clinical interview for DSM-V. Healthy controls will be matched to the patient sample.
Sampling Method: Non-Probability Sample
Enrollment: 102 (Actual)
Dates: Start 2021-05-03 (Actual); Primary Completion 2024-06-14 (Actual); Study Completion 2024-07-26 (Actual)

PRIMARY OUTCOMES:
Change in depression severity after the treatment phase | Up to 5 weekdays after the last iTBS treatment session
  Measured with the Montgomery Asberg Rating Scale (MARDS). Remission defined as MADRS score (range: 0 to 60) of less than or equal to 10. Response defined as a reduction of at least 50 percent from baseline in MADRS score.
Change in BPD severity after the treatment phase | Up to 5 weekdays after the last iTBS treatment session
  Measured by the Zanarini rating scale for BPD (Zan-BPD, range 0-36). Remission is defined as score of 9 or less. Response defined as a decrease from baseline in Zan-BPD score of at least 20 percent of the scoring range, i.e. a reduction of 8 points or more.
Changes in neural responses in an interoception task before the first and after the last treatment session | Up to 5 weekdays before the first and after the last treatment session
  Measured with functional magnetic resonance imaging (fMRI) while performing an interoception task
Changes in neural responses in a cognitive control task before the first and after the last treatment session | Up to 5 weekdays before the first and after the last treatment session
  Measured with functional magnetic resonance imaging (fMRI) while performing a cognitive control task
Changes in behavioral responses in an interoception task before the first and after the last treatment session | Up to 5 weekdays before the first and after the last treatment session
  Measured as performance in an interoception task during fMRI
Changes in behavioral responses in a cognitive control task before the first and after the last treatment session | Up to 5 weekdays before the first and after the last treatment session
  Measured as performance in a cognitive control task during fMRI
Changes in sleep staging over the treatment course | 2 days of baseline measurement before the first iTBS session, daily over the treatment course for 10 days
  electroencephalography (EEG)-based sleep staging measured with a headband device with accelerometer and pulseoximeter

SECONDARY OUTCOMES:
Changes in brain connectivity measures | Up to 5 weekdays before the first and after the last treatment session
  Structural and functional connectivity measured with MRI including graph measures
Changes in vigilance over the treatment course | Baseline immediately before the first iTBS session, daily over the treatment course for 10 days
  Vigilance measured by Psychomotor Vigilance Task (PVT)
Changes in symptom severity over treatment course | Baseline immediately before the first iTBS session, after 1 week of treatment, after 2 weeks of treatment, and at the follow-up 6 weeks after treatment
  Measured by the MADRS
Changes in self-reported symptom severity over treatment course and at follow-up | Baseline immediately before the first iTBS session, daily over the treatment course for 10 days, 6 weeks after last iTBS session at the follow-up
  measured by the Beck Depression Inventory (BDI-II)
Changes in Cortisol Awakening Response (CAR) from saliva concentrations | Up to 5 weekdays before the first and after the last treatment session
  3 measurements after awakening (0,20, and 40 minutes)
Changes in blood parameters | Before the first and after the last treatment session
  Pro- and anti-inflammatory cytokines, and growth factors
Association between changes induced by the Forecaster session and treatment outcome | Immediately before and after the forecaster iTBS session
  Changes in biomarkers before and after the forecaster iTBS session
Changes in self-reported BPD symptom severity over treatment course and at follow-up | Baseline immediately before the first iTBS session, daily over the treatment course for 10 days, 6 weeks after last iTBS session at follow-up
  Measured by the Borderline Symptom List (BSL-23) (range 0-4)
Changes in BPD symptom severity over treatment course and at follow-up | Baseline immediately before the first iTBS session, after 1 week of treatment, and after 2 weeks of treatment
  Measured by Zan-BPD
Changes in food craving | Up to 5 weekdays before the first and after the last treatment session
  Measured by a behavioral food craving task

CONTACTS AND LOCATIONS:
Overall Officials: René Hurlemann, Prof., Principal Investigator — Department of Psychiatry, University of Oldenburg; Dirk Scheele, Dr., Principal Investigator — Department of Psychiatry, University of Oldenburg; Christina Mueller, M.Sc., Study Director — Department of Psychiatry, University of Oldenburg; Marc Onken, M.Sc., Study Director — Department of Psychiatry, University of Oldenburg
Locations (1):
- Department of Psychiatry, University of Oldenburg, Bad Zwischenahn, Germany

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Blumberger DM, Vila-Rodriguez F, Thorpe KE, Feffer K, Noda Y, Giacobbe P, Knyahnytska Y, Kennedy SH, Lam RW, Daskalakis ZJ, Downar J. Effectiveness of theta burst versus high-frequency repetitive transcranial magnetic stimulation in patients with depression (THREE-D): a randomised non-inferiority trial. Lancet. 2018 Apr 28;391(10131):1683-1692. doi: 10.1016/S0140-6736(18)30295-2. Epub 2018 Apr 26. PMID 29726344
- [Background] Franzen PL, Buysse DJ. Sleep disturbances and depression: risk relationships for subsequent depression and therapeutic implications. Dialogues Clin Neurosci. 2008;10(4):473-81. doi: 10.31887/DCNS.2008.10.4/plfranzen. PMID 19170404
- [Background] Mutz J, Vipulananthan V, Carter B, Hurlemann R, Fu CHY, Young AH. Comparative efficacy and acceptability of non-surgical brain stimulation for the acute treatment of major depressive episodes in adults: systematic review and network meta-analysis. BMJ. 2019 Mar 27;364:l1079. doi: 10.1136/bmj.l1079. PMID 30917990
- [Background] Rock PL, Roiser JP, Riedel WJ, Blackwell AD. Cognitive impairment in depression: a systematic review and meta-analysis. Psychol Med. 2014 Jul;44(10):2029-40. doi: 10.1017/S0033291713002535. Epub 2013 Oct 29. PMID 24168753
- [Background] Tsuno N, Besset A, Ritchie K. Sleep and depression. J Clin Psychiatry. 2005 Oct;66(10):1254-69. doi: 10.4088/jcp.v66n1008. PMID 16259539